CLINICAL TRIAL: NCT06765590
Title: A Randomized, Open-label, Single-dose, Two-period, Two-way Crossover Bioequivalence Study of Paclitaxel for Injection (Albumin Bound) in Subjects With Breast Cancer
Brief Title: Bioequivalence Study of Paclitaxel for Injection (Albumin Bound) in Subjects With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: The First Hospital of Jilin University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Chongqing Traditional Chinese Medicine Hospital (Other); The First Affiliated Hospital of Henan University of Science and Technology (Other); Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HY-PA023-001
Record Dates: First submitted 2024-12-23; First posted 2025-01-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test preparation T: Paclitaxel for injection (albumin-bound) (Experimental)
  Interventions: Drug: T, 260 mg/m2, paclitaxel for injection (albumin-bound)
- Reference Preparation R: Paclitaxel (albumin-bound) for injection (Trade name: ABRAXANE) (Experimental)
  Interventions: Drug: R, 260 mg/m2, paclitaxel for injection (albumin bound).

INTERVENTIONS:
Drug: T, 260 mg/m2, paclitaxel for injection (albumin-bound) — T, 260 mg/m2, paclitaxel for injection (albumin-bound)
  Arms: Test preparation T: Paclitaxel for injection (albumin-bound)
Drug: R, 260 mg/m2, paclitaxel for injection (albumin bound). — R, 260 mg/m2, paclitaxel for injection (albumin bound).
  Arms: Reference Preparation R: Paclitaxel (albumin-bound) for injection (Trade name: ABRAXANE)

SUMMARY:
This study was a multicenter, randomized, open, single-dose, two-cycle, two-cross-dosing human bioequivalence trial designed to evaluate the bioequivalence of tested and reference preparations in breast cancer subjects.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, open, single-dose, two-cycle, two-cross-dosing human bioequivalence trial designed to evaluate the bioequivalence of tested and reference preparations in breast cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in the study and sign the informed consent forms (ICFs);
2. Patients with breast cancer confirmed by histopathology and/or cytology who meet one of the following conditions: ① with metastatic breast cancer that does not respond to combination chemotherapy or recurrent breast cancer within 6 months after adjuvant chemotherapy, and an anthracycline anticancer drug should be used in the previous chemotherapy unless clinically contraindicated; ② investigators determine that subjects are candidates for albumin-bound paclitaxel by reference to the treatment guidelines (NCCN Guidelines and CSCO Guidelines for breast cancer);
3. Aged 18-75 years old (both inclusive), males or females; body mass index (BMI) ≥17 (BMI = weight (kg)/height (m2));
4. The ECOG score is 0-2;
5. The expected survival time is ≥3 months;
6. Subjects have no plans to become pregnant and voluntarily use non-pharmacologic contraception (such as total abstinence, condom, contraceptive ring, vasectomy, etc.) or other highly effective contraceptive methods, and have no plans to donate eggs or sperm throughout the trial and within 6 months after the last dose;
7. Subjects with the laboratory test results as follows: hemoglobin (Hb) ≥80 g/L (no blood transfusion within 14 days), absolute neutrophil count (ANC) ≥1.5 * 109/L, platelet count (PLT) ≥100 * 109/L; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times the upper limit of normal value (for patients without liver metastasis) or ≤5 times the upper limit of normal value (for patients with liver metastasis); total bilirubin (TBIL) ≤1.5 times the upper limit of normal value (for patients without liver metastasis) or ≤3 times the upper limit of normal value (for patients with liver metastasis); serum creatinine clearance ≥60 mL/min [formula: Ccr: (140 - age) * body weight (kg) * 0.85 (if female)/0.818 * Scr (μmol/L)]; international normalized ratio (INR) ≤1.5 times the upper limit of normal value;
8. Subjects are able to communicate well with the investigator and understand and comply with the requirements of the study.

Exclusion Criteria:

1. Subjects with allergic constitution (excluding mild asymptomatic seasonal allergies), or who are known (or suspected) to be allergic to or have a specific reaction to the active ingredient paclitaxel or excipients, albumin;
2. Subjects who have received radiotherapy, chemotherapy, immunotherapy and endocrinotherapy within 4 weeks before the administration of the investigational drug and still respond to the treatment;
3. Subjects who have suffered from serious illness of cardio-cerebral vascular system, lung, liver, kidney, gastrointestinal tract, endocrine system, immune system, skin, musculoskeletal system and nervous system or psychiatric disorders within 3 months before screening and are considered unsuitable for enrollment by the investigator;
4. Subjects who have undergone major surgery or suffered from fracture within 4 weeks prior to screening, or plan to undergo major surgery during the study;
5. Subjects who have received treatment with other investigational drugs within 4 weeks before the study;
6. Subjects who have used substrates, inducers or inhibitors of CYP2C8 or CYP3A4 enzymes (including but not limited to ketoconazole and other imidazole antifungal agents, verapamil, diazepam, quinidine, dexamethasone, cyclosporine, teniposide, etoposide, vincristine, testosterone, 17-α diethylstilbestrol, retinoic acid, quercetin, erythromycin, fluoxetine, gemfibrozil, cimetidine, ritonavir, saquinavir, indinavir, nelfinavir, rifampicin, carbamazepine, phenytoin, efavirenz, nevirapine, etc.) in concomitant medications within 4 weeks prior to the first dose of the investigational drug or fail to suspend medications during the study (except for stable dosing at steady state, i.e. the dosing regimen remains unchanged);
7. Subjects who have consumed special diet (foods that affect the activity of CYP3A4 or CYP2C8 enzyme, such as grapefruit, pomelo, mango, etc.), exercised vigorously or with other factors that may affect drug absorption, distribution, metabolism and excretion within 48 hours before the administration of the investigational drug;
8. Subjects who have received therapy with the granulocyte colony-stimulating factor (G-CSF) within 2 weeks before screening;
9. Subjects with grade 2 or higher sensory neuropathy/peripheral neuropathy at screening;
10. Subjects who have experienced myocardial infarction (within 6 months before the study), severe or unstable angina, and grade III-IV heart failure according to the New York Heart Association (NYHA) Classification, or underwent coronary or peripheral artery bypass grafting;
11. Subjects with poorly controlled hypertension (with the systolic blood pressure of >160 mmHg and/or diastolic blood pressure of >100 mmHg under regular medication);
12. Subjects who have bleeding tendency or are receiving thrombolytic or anticoagulant therapy or have donated or lost more than 400 mL of blood within 3 months before the administration of the investigational drug;
13. Subjects with clinically significant 12-lead ECG abnormalities, who are considered unsuitable for enrollment by the investigator;
14. Subjects with a history of alcohol (drinking more than 14 units of alcohol per week within 6 months prior to the first dose: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), drug abuse (using narcotic drugs or psychotropic drugs for non-medical purposes) or addiction to drugs, who smoked more than 5 cigarettes per day within 3 months prior to screening, or who could not stop smoking or drinking during the period from signing the ICFs to completing the bioequivalence study;
15. Subjects with positive results of hepatitis B surface antigen (HBsAg), HBV DNA, hepatitis C core antibody (HCV-cAg), HCV RNA, HIV antibody, treponema pallidum antibody, or rapid plasma reagin (RPR) test;
16. Pregnant or lactating women;
17. Other conditions judged inappropriate for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-01-10 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Maximum observed concentration of paclitaxel (Cmax) | Predose: 0 hours; Post-infusion: 0.25 hours, 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours.
Area under the concentration-time curve from time zero to infinite time of paclitaxel (AUC 0-inf) | Predose: 0 hours; Post-infusion: 0.25 hours, 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours.
Area under the concentration-time curve from time zero to the last time of paclitaxel (AUC 0-t) | Predose: 0 hours; Post-infusion: 0.25 hours, 0.5 hours, 0.75 hours, 1 hour, 1.5 hours, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 36 hours, 48 hours, and 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated hospital of Hennan University of Science & Technology, Luoyang, Henan, China

IPD SHARING:
Plan to Share IPD: No